CLINICAL TRIAL: NCT05748366
Title: Ultrasound Guided Serratus Anterior Plane Block Versus Standard Therapy for Analgesic Relief of Rib Fractures in the Emergency Department
Brief Title: Ultrasound Guided Serratus Anterior Plane Block for Rib Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Daniel Kreider, Associate Director of Emergency Ultrasound, Principal Investigator, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-2023-30
Record Dates: First submitted 2023-02-14; First posted 2023-02-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Rib Fracture Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Serratus Anterior Plane Block (Experimental): Subjects will undergo serratus anterior plane block, in addition to standard of care analgesic medications at the discretion of the treatment team.
  Interventions: Procedure: Serratus Anterior Plane Block (SAPB); Drug: Standard Analgesic Medications
- Standard Analgesic Medications (Active Comparator): Subjects will receive standard of care analgesic medications at the discretion of the treatment team.
  Interventions: Drug: Standard Analgesic Medications

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block (SAPB) — The ultrasound-guided serratus anterior plane block (SAPB) will be performed in a manner previously described in published medical literature. Patients will be consented and monitored. Bupivacaine 0.5% (5 mg/ml) diluted to 30-40 ml will be used in a dose not to exceed 2 mg/kg. The serratus anterior fascial plane will be identified in the 4th/5th intercostal space. The needle will be advanced under real-time ultrasound guidance targeting the superficial serratus anterior fascial plane. The procedure assistant will inject small volumes to hydrodissect the muscle bellies evenly under direct visualization, indicating local anesthetic spread within the fascial plane. Anesthetic will then be injected in 5 ml increments and the needle will be removed. Patient will be continuously monitored on telemetry and pulse-oximetry. Reassessment of the patient will continue for 30 minutes to monitor for signs of local anesthetic systemic toxicity.
  Other Names: SAPB
  Arms: Serratus Anterior Plane Block
Drug: Standard Analgesic Medications — Analgesic medications will be administered via the intravenous, intramuscular or oral route at the discretion of the medical treatment team.

SUMMARY:
This study is a single center, randomized controlled trial examining the effect of serratus anterior plane block (SAPB) on pain, PIC scores and other clinical outcomes in emergency department patients with multiple rib fractures in comparison to the use of analgesic medication alone.

Objectives

1. Compare SAPB performed in the ED setting to analgesic medication alone with regard to pain, respiratory status and PIC score of patients with multiple rib fractures.
2. Assess the safety and feasibility of performing ultrasound-guided SAPB in the ED.
3. Evaluate outcomes of patients receiving the SAPB in the ED including amount of analgesic medications used, level of care required, need for upgrading level of care, and length of stay.

DETAILED DESCRIPTION:
Background Rib fractures are a common injury encountered in the emergency department (ED) affecting an estimated 10% of all trauma patients. They are associated with significant morbidity and mortality, especially in elderly patients. Rib fractures are the leading indication for intensive care unit (ICU) admission in patients with traumatic injuries to the thorax, accounting for approximately 42% of patients who require critical care in trauma. Secondary complications from rib fractures include atelectasis, pneumonia, and acute respiratory distress syndrome. These complications are often attributed to a relative respiratory functional deficit secondary to pain which limits adequate inspiratory capacity and coughing; therefore, the management of acute rib fractures has largely been focused on controlling pain. The most common method of pain control employed in the ED has historically been the use of a multimodal analgesic approach which includes opioids, acetaminophen, and NSAIDS. Opioids confer additional risks which include respiratory depression, suppressed cough reflex, delirium, nausea, constipation, and the potential for addiction.

Ultrasound-guided serratus anterior plane block (SAPB) is an alternative method of pain control that utilizes targeted delivery of a local anesthetic agent in the serratus anterior fascial plane. This method was first described in 2013 and has been well described for the treatment of pain associated with thoracic surgical procedures, including those of the breast and chest wall. The SAPB has also been demonstrated to provide analgesic relief of pain associated with rib fractures and other blunt chest-wall traumatic injuries.

Over recent years, the SAPB technique has been gaining popularity due to its efficacy, relative ease of performance, and favorable side effect profile. This ultrasound guided technique uses a high frequency linear ultrasound transducer to identify the serratus anterior fascial planes, latissimus dorsi muscle, ribs, and pleural space. The intended target is the superficial serratus anterior fascial plane, which is bordered by the latissimus dorsi muscle posteriorly and the pectoralis muscles anteriorly. This fascial plane houses the lateral cutaneous branches of the intercostal nerves and a plane block of the superior facial plane has also been postulated to provide analgesia in the distribution of the long thoracic and thoracodorsal nerves. The block primarily works at the level of T2-T9, and previous literature has suggested that the SAPB works best for anterolateral rib fractures. The SAPB has a relatively safe side effect profile. Major complications include pneumothorax and local anesthetic systemic toxicity (LAST); however, the incidence of adverse events following SAPB performed in the ED has been low in previous studies.

Point of care ultrasound (POCUS) for procedural guidance is commonly employed by emergency physicians in daily clinical practice. Several retrospective and case-series studies have demonstrated the efficacy, feasibility, and safety of SAPB in the ED when performed by trained ED physicians. Studies like those performed by Diwan et al. and Kring et al. have demonstrated improved pain scores and decreased opioid consumption following SAPB. Despite this, to date, there has only been one published randomized controlled trial comparing the analgesic effects of SAPB versus opioid pain medication. More data is needed to further evaluate the analgesic effect of ED performed SAPB and the outcome of patients who present with acute rib fractures.

The Pain, Inspiratory capacity, and Cough (PIC) score is a tool currently utilized in blunt chest trauma cases at WellSpan York Hospital to guide inpatient management and predict the need for escalating care. This ten-point scoring tool accounts for the patient's pain level (mild/moderate/severe), inspiratory capacity (percent predicted value), and cough effort, with a goal score of >8. Inspiratory capacity and cough effort are often directly related to the level of pain a patient is experiencing, therefore, improving rib fracture pain through SAPB may improve PIC scores and help reduce the need for intensive care unit (ICU) level care. Additionally, analgesic relief with SAPB should decrease opioid consumption and its associated risks in the immediate period following rib fractures.

The goal of this study is to examine the effect of ED-performed SAPB on pain, PIC scores and other clinical outcomes in patients with multiple rib fractures in comparison to the use of analgesic medication alone.

Objectives

1. Compare SAPB performed in the ED setting to analgesic medication alone with regard to pain, respiratory status and PIC score of patients with multiple rib fractures.
2. Assess the safety and feasibility of performing ultrasound-guided SAPB in the ED.
3. Evaluate outcomes of patients receiving the SAPB in the ED including amount of analgesic medications used, level of care required, need for upgrading level of care, and length of stay.

Outcomes: See subsequent entries.

Research methods

Study design This will be a randomized, controlled, superiority trial consisting of adult patients presenting to the WellSpan York Hospital ED with >1 unilateral rib fracture on either x-ray or CT imaging. Screening for potential subjects will be conducted by ED staff working clinically, as well as ultrasound/procedure emergency medicine residents and US fellows/faculty on "scanning shifts." Informed consent will be obtained by a member of the study team prior to data collection or study procedures. Patients enrolled in the study will be randomized to one of two groups. Group 1 (control) will receive standard multimodal pain control as deemed appropriate by the treating physician. Group 2 (intervention) will receive the SAPB according to the attached protocol, as well as standard multimodal analgesia per standard of care. It should be emphasized that patients in group 2 will still receive standard multimodal pain medication at the discretion of the treating physician if the SAPB is not providing adequate analgesic relief. Both SAPB and analgesic medications fall within the current standard of care for pain management in rib fractures.

A point-of-care (POC) ultrasound will be performed by an ED attending, fellow or resident under the supervision of an emergency physician accredited in ultrasound-guided SAPB. Clinical and demographic data, including the number and location of rib fractures, procedural details, and initial pain/PIC scores will be documented at the bedside. Ultrasound images will be recorded via the usual ultrasound archival software and undergo the standard QA process used for all POC US studies performed in the ED. ED residents/fellows/attendings participating in this study will be trained on study protocols by accredited staff prior to participation in consent, ultrasonography and data collection.

Additional follow up data will be collected via a phone call at 1 week and a review of the electronic medical record at 30 days. All research data will be documented on standardized data collection forms.

Study population and recruitment Study population will include ED patients over the age of 18 identified with rib fractures on x-ray or CT imaging. Patients will be seen initially by the treating physician and receive the usual standard of care. If rib fractures are identified, the treating physician will contact a member of the study team to assess eligibility, discuss the study with the patient and/or the legally authorized representative (LAR) and obtain consent. The POC ultrasound procedure may be performed by a physician member of the study team or another credentialed emergency physician.

Inclusion/exclusion criteria: See subsequent entries.

Role of subjects Study participants will receive standard treatment at the discretion of the treating physician or advanced practice provider. The patient's decision to participate in this study will not directly affect their care in the ED. The treating provider will not necessarily be blinded to the treatment provided as they will need to perform the SAPB if the patient is randomized to the interventional group 2.

Research procedures Screening for inclusion in this study will occur in the ED as outlined above. Informed consent will be given to eligible patients/LARs for review. Written informed consent will be obtained prior to randomization to treatment vs control group. If randomized to the control group, patients will sign a separate procedure consent form for SAPB.

Each patient will be assigned a study ID number at the time of enrollment and a linking document will be maintained. Once data collection is complete, forms will be de-identified by the removal of the patient's name/MRN/FIN/identifying information.

Randomization will be determined by pre-filled, numbered study folders available in the ED at the start of the study. Each enrolled subject will be randomized based on the contents of the study folder labeled with their corresponding study ID number.

Of note, subjects initially assigned to group 1 (control) are eligible to crossover and undergo SABP if their pain is inadequately controlled 2 hours post-randomization or later. This option will be left up to shared decision-making between the treating physicians and patient.

All patients undergoing SABP will be additionally consented specifically for the medical procedure per usual ED standard of care.

Ultrasound/Procedural technique: Please see later fields.

Data analysis and sample size calculations Descriptive statistics will be reported as means/medians with standard deviation/interquartile range for continuous variables and proportions with percentages for categorical variables. Differences in continuous outcome variables between study groups will be compared via Student T-test for parametric data and Mann-Whitney U test for non-parametric data with associated 95% confidence intervals. Differences in dichotomous variables between groups will be compared via chi-squared or Fisher's exact tests, as appropriate. Primary analysis will be conducted on an intention to treat basis; however, given the potential for cross-over, per protocol sensitivity analysis is also planned. Interrater reliability for follow up data collection from the medical record will be assessed via Cohen's kappa. p<0.05 will be considered statistically significant. Statistical analysis will be performed using SPSS software (IBM, Armonk, NY).

Power calculations are based on prior published literature and local data on patients admitted to WellSpan York Hospital with rib fractures over the past year. We assume a baseline pain VAS mean=7.7/SD=2.2, an expected mean 2-hour pain VAS change difference between study groups of 2.5 and a margin of superiority of 1.0. Allowing for 5-10% attrition, we plan to enroll a total of 60 subjects (30 per arm, randomized 1:1) to achieve 80% power at alpha=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* >1 Unilateral, acute rib fractures diagnosed on x-ray or CT imaging
* Patient presenting to the WellSpan York Hospital ED
* Patient requiring IV analgesia or oral opioid to control pain related to rib fractures

Exclusion Criteria:

* Age <18 years
* Inability to provide informed consent
* Allergy to local anesthesia
* Subsequent visit for rib fractures
* Patients taken emergently to the OR or discharged from the ED
* Significant distracting injuries/polytrauma that would not be expected to be responsive to analgesia from SAPB and confound pain scores, i.e. long bone fractures, intraabdominal injuries, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Score (VAS) at 2 hours | 2 hours
  Change in pain score on a visual analog scale (VAS) at 2 hours following randomization to ultrasound guided SAPB or analgesic medication only.

SECONDARY OUTCOMES:
Pain Score | 4 hours, 6 hours, 8 hours, and 12 hours following randomization
  Numerical pain score (0-10 scale) at 4 hours, 6 hours, 8 hours, and 12 hours following randomization
Pain/Inspiratory Effort/Cough (PIC) Score | 4 hours, 6 hours, 8 hours, and 12 hours following randomization
  PIC score (0-10 scale) at 4 hours, 6 hours, 8 hours, and 12 hours following
Morphine Milligrams Equivalent (MME) | 2 hours, 4 hours, 6 hours, 8 hours and 12 hours following randomization
  Morphine milligram equivalents (MME) of analgesia consumed at 2 hours, 4 hours, 6 hours, 8 hours and 12 hours following randomization
Length of Stay (hours) | During index hospitalization following randomization
  Emergency department, hospital and ICU lengths of stay
Rate of ICU Utilization | From date of randomization until the date of discharge from the hospital or death from any cause, whichever came first, assessed up to 100 months
  Hospitalization at ICU level care or upgrade to ICU level care during index hospitalization
Rate of Crossover | From date/time of randomization until the date/time of departure from the ED or death from any cause, whichever came first, assessed up to 24 hours
  Crossover from standard analgesic medication arm to the serratus anterior plane block arm due to inadequate pain control.

OTHER OUTCOMES:
Safety Outcomes | 30 days
  Adverse outcomes related to serratus anterior plane block, including systemic toxicity, infection, pneumothorax, nerve injury or other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Kreider, MD, Principal Investigator — WellSpan Health
Locations (1):
- Wellspan Health York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Southgate SJ, River GF, Herbst MK. Ultrasound-Guided Serratus Anterior Blocks. 2024 Feb 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK538476/ PMID 30860711
- [Background] Terry SM, Shoff KA, Sharrah ML. Improving Blunt Chest Wall Injury Outcomes: Introducing the PIC Score. J Trauma Nurs. 2021 Nov-Dec 01;28(6):386-394. doi: 10.1097/JTN.0000000000000618. PMID 34766933
- [Background] Bass GA, Stephen C, Forssten MP, Bailey JA, Mohseni S, Cao Y, Chreiman K, Duffy C, Seamon MJ, Cannon JW, Martin ND. Admission Triage With Pain, Inspiratory Effort, Cough Score can Predict Critical Care Utilization and Length of Stay in Isolated Chest Wall Injury. J Surg Res. 2022 Sep;277:310-318. doi: 10.1016/j.jss.2022.04.001. Epub 2022 May 6. PMID 35533604
- [Background] Witt CE, Bulger EM. Comprehensive approach to the management of the patient with multiple rib fractures: a review and introduction of a bundled rib fracture management protocol. Trauma Surg Acute Care Open. 2017 Jan 5;2(1):e000064. doi: 10.1136/tsaco-2016-000064. eCollection 2017. PMID 29766081
- [Background] Schnekenburger M, Mathew J, Fitzgerald M, Hendel S, Sekandarzad MW, Mitra B. Regional anaesthesia for rib fractures: A pilot study of serratus anterior plane block. Emerg Med Australas. 2021 Oct;33(5):788-793. doi: 10.1111/1742-6723.13724. Epub 2021 Jan 29. PMID 33511786
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Nair A, Diwan S. Efficacy of Ultrasound-Guided Serratus Anterior Plane Block for Managing Pain Due to Multiple Rib Fractures: A Scoping Review. Cureus. 2022 Jan 17;14(1):e21322. doi: 10.7759/cureus.21322. eCollection 2022 Jan. PMID 35186581
- [Background] Davis K, Connor X. Single injection serratus anterior plane blocks for traumatic rib fractures. A good start but a missed opportunity. Am J Emerg Med. 2021 Dec;50:810. doi: 10.1016/j.ajem.2021.03.045. Epub 2021 Mar 14. No abstract available. PMID 33745771
- [Background] Diwan S, Nair A. A retrospective study comparing analgesic efficacy of ultrasound-guided serratus anterior plane block versus intravenous fentanyl infusion in patients with multiple rib fractures. J Anaesthesiol Clin Pharmacol. 2021 Jul-Sep;37(3):411-415. doi: 10.4103/joacp.JOACP_349_19. Epub 2021 Oct 12. PMID 34759553
- [Background] Kring RM, Mackenzie DC, Wilson CN, Rappold JF, Strout TD, Croft PE. Ultrasound-Guided Serratus Anterior Plane Block (SAPB) Improves Pain Control in Patients With Rib Fractures. J Ultrasound Med. 2022 Nov;41(11):2695-2701. doi: 10.1002/jum.15953. Epub 2022 Feb 2. PMID 35106815
- [Background] Lin J, Hoffman T, Badashova K, Motov S, Haines L. Serratus Anterior Plane Block in the Emergency Department: A Case Series. Clin Pract Cases Emerg Med. 2020 Jan 21;4(1):21-25. doi: 10.5811/cpcem.2019.11.44946. eCollection 2020 Feb. PMID 32064417
- [Background] Paul S, Bhoi SK, Sinha TP, Kumar G. Ultrasound-Guided Serratus Anterior Plane Block for Rib Fracture-Associated Pain Management in Emergency Department. J Emerg Trauma Shock. 2020 Jul-Sep;13(3):208-212. doi: 10.4103/JETS.JETS_155_19. Epub 2020 Sep 18. PMID 33304071
- [Background] Teksen S, Oksuz G, Oksuz H, Sayan M, Arslan M, Urfalioglu A, Gisi G, Bilal B. Analgesic efficacy of the serratus anterior plane block in rib fractures pain: A randomized controlled trial. Am J Emerg Med. 2021 Mar;41:16-20. doi: 10.1016/j.ajem.2020.12.041. Epub 2020 Dec 23. PMID 33383266
- [Background] Kelly AM. The minimum clinically significant difference in visual analogue scale pain score does not differ with severity of pain. Emerg Med J. 2001 May;18(3):205-7. doi: 10.1136/emj.18.3.205. PMID 11354213
- [Background] Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov;5(11):1086-90. doi: 10.1111/j.1553-2712.1998.tb02667.x. PMID 9835471